CLINICAL TRIAL: NCT04241133
Title: The UnProcessed Pantry Project (UP3): A Novel Approach to Improving Dietary Quality for Low-Income Adults Served by Rural Food Pantries
Brief Title: The UnProcessed Pantry Project (UP3)
Acronym: UP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: Center for American Indian and Rural Health Equity (Other); Gallatin Valley Food Bank (Other); Livingston Food Resource Center (Other); Bozeman Deaconess Health Group (Other); Gallatin City-County Health Department (Other); Helena Food Share (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CBS122118
Record Dates: First submitted 2019-09-26; First posted 2020-01-27 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Diet, Healthy; Diet Habit; Disease, Chronic; Health Behavior; Rural Health
MeSH Terms: conditions — Feeding Behavior; Chronic Disease; Health Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to an intervention group or control group (nonrandomized).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A 12 week pilot trial will be conducted at two rural food pantries in Montana with 40 low-income adults to measure within-participant changes over time. The study will provide the initial investigation of the extent to which UP3 will improve overall dietary quality as measured by the Healthy Eating Index-2015 (HEI) compared to baseline. Psychosocial factors will be measured to understand changes in knowledge, attitudes, and perceptions about processed foods. Data on biomarkers of health (i.e., weight, systolic blood pressure, HbA1c, fasting lipid panel) will be collected to assess the feasibility of measuring potential short-term health effects of UP3.
  Interventions: Behavioral: The UnProcessed Pantry Project (UP3)
- Control Group (No Intervention): 20 separate participants from a different food pantry will be enrolled into a control group. The control group will be assessed at baseline and 12 weeks for dietary intake, height, weight, waist circumference, food security, demographics, and psychosocial factors.

INTERVENTIONS:
Behavioral: The UnProcessed Pantry Project (UP3) — UP3 uses the Social-Ecological Model to target multiple levels, including the food supply in the rural study location (community level), the food environment at the food pantry (environmental level), and participant dietary intake (individual level). It is hypothesized that UP3 will improve access to minimally processed foods and decrease access to ultra-processed foods at the food pantry, which will improve overall dietary quality of individuals as measured by the Healthy Eating Index-2015 compared to baseline and to the control group. Demographic and food security data will characterize the population. Psychosocial factors will be collected to understand changes in knowledge, attitudes, and perceptions about processed foods. Biomarkers of health data (i.e., weight, systolic blood pressure, HbA1c, fasting lipid panel) will be collected to determine the feasibility of measuring potential short-term health effects alongside UP3.
  Arms: Experimental Group

SUMMARY:
There is a need to develop evidence-based interventions that rural food pantries can use to limit the distribution and intake of ultra-processed foods and promote the distribution and intake of minimally processed foods in the food environment and among low-income populations to promote better dietary quality and health outcomes. This research project, The UnProcessed Pantry Project (UP3): A Novel Approach to Improving Dietary Quality for Low-Income Adults Served by Rural Food Pantries, uses the Social-Ecological Model to target multiple levels, including the food supply in the rural study location (community level), the food environment at the food pantry (environmental level), and participant dietary intake (individual level). Aim 1 will adapt evidence-based strategies to inform UP3. UP3 will improve dietary quality by influencing the food supply through organization-wide nutrition policies, modifying the food environment with minimally processed foods and nudges, and changing participant dietary intake through experiential nutrition education. The UP3 pilot study will be conducted during Aim 2 with 40 participants served by two rural food pantries in Montana. The purpose of the pilot study is to investigate potential short-term effects on nutrient intake and dietary quality (primary outcome), assess acceptability of UP3 among participants, and evaluate feasibility in rural food pantry environments. It is hypothesized that UP3 will improve access to minimally processed foods and decrease access to ultra-processed foods at the food pantry, which will improve overall dietary quality of individuals as measured by the Healthy Eating Index-2015 compared to baseline and to the control group. Demographic and food security data will characterize the population. Psychosocial factors will be collected to understand changes in knowledge, attitudes, and perceptions about processed foods. Biomarkers of health data (i.e., weight, systolic blood pressure, HbA1c, fasting lipid panel) will be collected to determine the feasibility of measuring potential short-term health effects alongside UP3. A control group of 20 participants at a rural food pantry will be used to assess dietary intake, psychosocial factors, height, and weight. Aim 3 will tailor UP3 for a scalable intervention suited for an R01 grant application to conduct a randomized controlled trial (RCT). UP3 is positioned to demonstrate the positive effects of limiting processed foods and increasing unprocessed and minimally processed foods on diets and, potentially, health among low-income populations. The short-term goals of this research are to develop an adaptable and scalable intervention suitable for rural food pantries serving low-income populations, as well as potentially contribute to a knowledge base around potential short-term effects of the minimally processed foods diet on dietary quality and health risks in those populations. The longer-term goals are to test the efficacy of the intervention in an RCT and then disseminate the approach to be integrated into rural food pantries serving low-income populations with the goal of decreasing health risks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above
* Attend 1 of the food pantry sites
* Ability to attend intervention and measurement activities
* Chronic disease risk

Exclusion Criteria:

* Pregnancy
* Unstable vital signs
* Food allergy as measured by baseline screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Byker Shanks, PhD RDN, Principal Investigator — Montana State University
Locations (1):
- Montana State University Health Sciences Building, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
Each participant will be assigned a code. The code will be connected with the participant's name and contact information on a separate Excel spreadsheet that is saved and stored securely on the PI's computer. Only coded IPD will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Only available on a secure server and file to study staff when needed for planning and analysis.
Access Criteria: A researcher with IRB approval

REFERENCES:
- [Background] Byker Shanks C, Weinmann E, Holder J, McCormick M, Parks CA, Vanderwood K, Coburn C, Johnson N, Yaroch AL. The UnProcessed Pantry Project Framework to Address Nutrition in the Emergency Food System. Am J Public Health. 2019 Oct;109(10):1368-1370. doi: 10.2105/AJPH.2019.305292. No abstract available. PMID 31483716
- [Background] Byker Shanks C, Webber E, Larison L, Wytcherley B. The translational implications of applying multiple measures to evaluate the nutrient quality of the food supply: a case study of two food pantries in Montana. Transl Behav Med. 2020 Dec 31;10(6):1367-1381. doi: 10.1093/tbm/ibaa108. PMID 33421084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: UP3 participants who accessed one of the two food pantry sites were asked to participate in UP3 through flyers and on-site recruitment from December 2019 to January 2020. First participant enrolled on January 24, 2020. Control group participants were recruited through flyers and on-site recruitment in March 2020 from another food pantry site.
Groups:
- Experimental Group: For a 12 week pilot trial, 44 adults enrolled in the UP3 intervention and within-participant changes were measured over time. The UnProcessed Pantry Project (UP3): UP3 uses the Social-Ecological Model to target multiple levels, including the food supply in the rural study location (community level), the food environment at the food pantry (environmental level), and participant dietary intake (individual level). It was hypothesized that UP3 will improve access to minimally processed foods and decrease access to ultra-processed foods at the food pantry, which will improve overall dietary quality of individuals as measured by the Healthy Eating Index-2015 compared to baseline and to the control group.
- Control Group: 34 participants enrolled from a different food pantry were enrolled into a control group. The post assessment was cancelled due to COVID-19 precautions.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 44 | 34
Completed | 30 | 0
Not Completed | 14 | 34
Not completed — COVID19 Precautions | 14 | 34

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: A 12 week pilot trial was conducted at two rural food pantries in Montana with low-income adults to measure within-participant changes over time. The UnProcessed Pantry Project (UP3): UP3 used the Social-Ecological Model to target multiple levels, including the food supply in the rural study location (community level), the food environment at the food pantry (environmental level), and participant dietary intake (individual level). It was hypothesized that UP3 will improve access to minimally processed foods and decrease access to ultra-processed foods at the food pantry, which would improve overall dietary quality of individuals as measured by the Healthy Eating Index-2015 compared to baseline and to the control group.
- Control Group: Participants from a different food pantry were be enrolled into a control group with no intervention.
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 44 | 34 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 28 | 64
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 18 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 43 | 32 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 1 | 1
  White | 40 | 29 | 69
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 34 | 78
Healthy Eating Index 2015 Scale [Mean (Standard Deviation); unit: units on a scale] — Data collected through Automated Self-Administered 24-hour dietary recall to calculate HEI-2015 scores. The scores range from 0 to 100, with higher scores reflecting greater adherence with dietary recommendations from the Dietary Guidelines for Americans. A score of 100 reflects high adherence and a score of 0 reflects no adherence.
  units on a scale | 47.14 (13.41) | 52.01 (10.45) | 49.58 (11.93)

OUTCOME MEASURES:

1. Primary Outcome: Dietary Quality Change
Description: The Healthy Eating Index-2015 scale was calculated from collected 24-hour dietary recall data collected using the ASA24 (Automated-Self Administered Recall System) a computerized dietary assessment tool. ata collected through Automated Self-Administered 24-hour dietary recall to calculate HEI-2015 scores. The scores range from 0 to 100, with higher scores reflecting greater adherence with dietary recommendations from the Dietary Guidelines for Americans. A score of 100 reflects high adherence and a score of 0 reflects no adherence.
Time Frame: Change from baseline dietary quality at 12 weeks
Population: Due to the onset of COVID19 at the same time of the post measure (simultaneous with stay at home orders), 14 participants did not complete the experimental group and the control group data was not collected.
Measure: Mean (Standard Deviation); unit: Change in HEI-2015 baseline to 12 weeks
Groups:
- Experimental Group: A 12 week pilot trial will be conducted at two rural food pantries in Montana with low-income adults to measure within-participant changes over time. The study will provide the initial investigation of the extent to which UP3 will improve overall dietary quality as measured by the Healthy Eating Index-2015 (HEI) compared to baseline. It is hypothesized that UP3 will improve access to minimally processed foods and decrease access to ultra-processed foods at the food pantry, which will improve overall dietary quality of individuals as measured by the Healthy Eating Index-2015 compared to baseline and to the control group.
- Control Group: Participants from a different food pantry will be enrolled into a control group. The primary outcome measure will be dietary intake. No intervention will be applied.
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 30 | 0
Change in HEI-2015 baseline to 12 weeks | 57.01 (13.94) |
Statistical Analysis 1: Comparison: Experimental Group; The experimental group was tested for significant difference in Healthy Eating Index 2015 (HEI-2015) scores at baseline and 12 weeks. SAS macros provided by the National Cancer Institute were used to compute HEI-2015 scores for each dietary recall at pre- (baseline) and post-intervention (12 weeks) using the Simple HEI Scoring Algorithm; Test type: Other — The experimental and control groups were not compared due to the inability to collect post data with the control group because of stay at home orders during the COVID-19 pandemic; p < 0.05, t-test, 2 sided — The reported P-value was calculated; The a priori threshold for statistical significance was P<0.05

ADVERSE EVENTS:
Time Frame: 12 weeks during intervention
Description: Serious Adverse Event Data was collected about health measures that may lead to inpatient hospitalization, including hemoglobin A1c, blood pressure, lipid panel, and weight change.
Groups:
- Control Group: Participants from a different food pantry were be enrolled into a control group with no intervention. The Healthy Eating Index-2015 was the primary outcome measure.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/34
Other Adverse Events (participants affected / at risk) | 0/44 | 0/34

LIMITATIONS AND CAVEATS:
Due to the onset of COVID19 at the same time of the post measure (simultaneous with stay at home orders), 14 participants did not complete the experimental group and the control group data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04241133/Prot_SAP_ICF_000.pdf